CLINICAL TRIAL: NCT05367336
Title: A Comparison of PLAtelet Response to Aspirin Between Emergency Department Patients With Chest Pain Receiving Fentanyl or Morphine (PLAAFM)
Brief Title: Platelet Reactivity With Fentanyl, Morphine, or no Narcotic
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: The study was halted prematurely due to difficulties in recruiting a sufficient number of participants. Despite efforts to enroll eligible individuals, the recruitment goals were not met, making it infeasible to continue the study as planned.
Sponsor: Corewell Health South (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: EGME#04-2021
Record Dates: First submitted 2021-09-23; First posted 2022-05-10 (Actual); Results first posted 2025-04-25 (Actual); Last update posted 2025-05-21 (Actual); Status verified 2025-05

CONDITIONS: Fentanyl; Platelet Reactivity
MeSH Terms: interventions — Morphine; Fentanyl

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Control (No Intervention): not receiving any narcotics
- Morphine (Experimental): the second group will be those receiving morphine
  Interventions: Drug: Morphine
- Fentanyl (Experimental): the 3rd group will be those receiving fentanyl
  Interventions: Drug: Fentanyl

INTERVENTIONS:
Drug: Morphine — second group will be receiving morphine
  Arms: Morphine
Drug: Fentanyl — third group receiving fentanyl
  Arms: Fentanyl

SUMMARY:
The goal is to determine whether fentanyl and morphine have similar effects in reducing aspirin's effect upon platelets in emergency department patients with chest discomfort. Morphine has been shown to worsen outcomes in heart attack patients due to reduction of oral anti-platelet agent effectiveness and so many providers have switches to using fentanyl. However, it is largely unknown whether fentanyl has similar effects.

DETAILED DESCRIPTION:
Patients presenting to the emergency department with chest discomfort who are being administered aspirin will be offered enrollment in this study. At the time of their zero and two hour troponin we will also draw platelet aggregration studies to determine the effects of aspirin upon platelets. Narcotic medicines slow the absorption of aspirin. Morphine has therefore been shown to decrease the effectiveness of aspirin. Many providers therefore use fentanyl instead, however little is known about the effects of fentanyl upon aspirin. We will therefore compare the platelet reactivity of patients receiving morphine, fentanyl, or no narcotics

ELIGIBILITY:
Inclusion Criteria:

* Adult Emergency Department patients undergoing 0 and 2 hour troponin testing
* administered aspirin within 30 minutes of the initial blood draw.
* patient presented via private vehicle
* provide informed consent
* over the age of 18

Exclusion Criteria:

* Patients not expected to get a 2 hour troponin;
* patients already on aspirin, clopidogrel, or stronger anti-coagulants;
* patients who arrived via EMS (Emergency Medical Services) given it can be difficult to find the run reports to determine whether patient received fentanyl in the pre-hospital period;
* pregnant patients;
* patients on chronic narcotics;
* patients already once enrolled in this study,
* inability to provide consent in English

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2022-08-31 (Actual); Primary Completion 2025-02-18 (Actual); Study Completion 2025-02-18 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Spectrum Health Lakeland, Saint Joseph, Michigan, United States

IPD SHARING:
Plan to Share IPD: No
Individual Participant Data (IPD) will not be shared due to the early termination of the study and the limited number of participants enrolled. Sharing IPD from a small sample size could compromise participant confidentiality and privacy. Ensuring the protection of participants' personal data is a priority, and the small number of participants increases the risk of identifying individuals.

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Control | Morphine | Fentanyl
Started | 13 | 2 | 6
Completed | 13 | 2 | 6
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Control | Morphine | Fentanyl | Total
Number analyzed (Participants) | 13 | 2 | 6 | 21
Age, Continuous [Mean (Standard Deviation); unit: years] | 54.67 (16.62) | 51.00 (14.14) | 56.17 (18.06) | 54.75 (16.08)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7 | 0 | 4 | 11
  Male | 6 | 2 | 2 | 10
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 2 | 0 | 1 | 3
  White | 10 | 2 | 5 | 17
  More than one race | 1 | 0 | 0 | 1
  Unknown or Not Reported | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 13 | 2 | 6 | 21

OUTCOME MEASURES:

1. Primary Outcome: Baseline Arachidonic Acid Maximum Aggregation (%) Result
Description: Arachidonic Acid Maximum Aggregation is assessed using light transmission aggregometry (LTA). This method involves adding arachidonic acid to platelet-rich plasma (PRP) and measuring the change in light transmittance as platelets aggregate. The maximum aggregation percentage is recorded as the highest point of aggregation observed during the test. From a clinical perspective, normal aggregation is considered 70% or higher and values below 70% may indicate platelet dysfunction or the influence of antiplatelet medications such as aspirin. In this study, the control group is expected to show a significant decrease in Arachidonic Acid Maximum Aggregation (%) from the baseline to the 2-hour mark. However, this decrease is anticipated to be smaller in the groups receiving morphine and fentanyl.
Time Frame: Baseline
Measure: Mean (Standard Deviation); unit: Arachidonic Acid Percent
Arm/Group | Control | Morphine | Fentanyl
Number analyzed (Participants) | 13 | 2 | 6
Arachidonic Acid Percent | 37.49 (35.14) | 39.00 (54.66) | 54.00 (41.56)

2. Primary Outcome: 2 Hour Arachidonic Acid Maximum Aggregation (%) Result
Description: as for outcome 1
Time Frame: 2 hours
Measure: Mean (Standard Deviation); unit: Arachidonic Acid Percent
Arm/Group | Control | Morphine | Fentanyl
Number analyzed (Participants) | 13 | 2 | 6
Arachidonic Acid Percent | 1.69 (0.56) | 1.00 (1.20) | 0.87 (1.63)

ADVERSE EVENTS:
Time Frame: Adverse event data were collected for up to 4 hours after arrival in the ED.
Arm/Group | Control | Morphine | Fentanyl
All-Cause Mortality (participants affected / at risk) | 0/13 | 0/2 | 0/6
Serious Adverse Events (participants affected / at risk) | 0/13 | 0/2 | 0/6
Other Adverse Events (participants affected / at risk) | 0/13 | 0/2 | 0/6

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2025-02-18): https://cdn.clinicaltrials.gov/large-docs/36/NCT05367336/Prot_SAP_000.pdf